CLINICAL TRIAL: NCT05641506
Title: An Open-label, Phase II Clinical Trial of of a Chinese Patent Medicine Yangzhengxiaoji Capsule to Improve the Adverse Reactions Nausea of Niraparib in in the First-line Maintenance Treatment in Advanced Epithelial Ovarian Cancer (EOC) Patients
Brief Title: A Chinese Patent Medicine Yangzhengxiaoji Capsule to Improve the Nausea of Niraparib in the Maintenance Treatment in Ovarian Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Guonan Zhang, Director, Head of Gynecologic Oncology Center, Sichuan Cancer Hospital and Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YONNY-2002-080
Record Dates: First submitted 2022-07-05; First posted 2022-12-07 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-11

CONDITIONS: Ovarian Cancer
Keywords: Niraparib, Ovarian Cancer,Nausea
MeSH Terms: conditions — Ovarian Neoplasms; Nausea | interventions — yangzheng xiaoji; niraparib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm (Experimental): Participants received Niraparib 200mg or 300mg QD PO continually combined with Yangzheng Xiaoji capsule， 0.36g*4 tid，28 days as one cycle，up to 3 cycles.
  Interventions: Drug: Yangzheng Xiaoji; Drug: Niraparib

INTERVENTIONS:
Drug: Yangzheng Xiaoji — Chinese patent medicine Yangzheng Xiaoji capsule， 0.36g*4 tid，28 days as one cycle，up to 3 cycles.
Drug: Niraparib — Niraparib 200 or 300mg* QD PO continually;
  *The starting dose of niraparib was individualized based on patients' bodyweight and baseline platelet count; 200 mg QD for Patients with baseline body weight <77 kg or platelets count <150,000/μL;300 mg QD for Patients with baseline body weight ≥77 kg and platelets count ≥150,000/μL.

SUMMARY:
This study is an open-label, single-Arm， phase II clinical trial of a Chinese Patent Medicine Yangzheng Xiaoji Capsule to improve the adverse reaction nausea of Niraparib in the first-line maintenance treatment in advanced epithelial ovarian cancer, fallopian tube cancer, and primary peritoneal cancer.

DETAILED DESCRIPTION:
This study will investigate a Chinese Patent Medicine Yangzheng Xiaoji Capsule improve the adverse reaction nausea of Niraparib in the first-line maintenance treatment in advanced EOC, who have previously received ≥ 3 cycles of prior combined bevacizumab chemotherapy and a complete or partial response with platinum-based chemotherapy.

Approximately 50 eligible subjects are planned to be enrolled, given Yangzheng Xiaoji Capsule and niraparib maintenance treatment.

The dosing regimen is:Niraparib 200mg QD combined with Yangzheng Xiaoji Capsule 0.36g*4 tid，28 days/cycle. Subjects will receive Niraparib plus Yangzheng Xiaoji Capsule up to 3 cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Sign a written informed consent form before conducting any research-related procedures;
2. Women aged 18 or above;
3. Ovarian cancer, fallopian tube cancer or primary peritoneal cancer diagnosed histologically can be treated with Niraparib after evaluation by clinicians;
4. Life expectancy > 3 months;
5. Patients' ECOG physical condition score is 0-1, KPS score is ≥70;
6. Patients received ≥ 3 cycles bevacizumab in combination within platinum-based chemotherapy
7. Good organ function, including:

   * Neutrophil count ≥ 1500/L
   * Platelet ≥ 100,000/L
   * Hemoglobin ≥10g/dL
   * Serum creatinine ≤1.5 times the upper limit of normal value, or creatinine clearance ≥60mL/min (according to Cockcroft-Gault Formula calculation)
   * Total bilirubin ≤1.5 times the upper limit of normal value or direct bilirubin ≤1.0 times the upper limit of normal value
   * AST and ALT ≤2.5 times the upper limit of normal value, and liver metastasis must be ≤5 times the upper limit of normal value.

7. No serious abnormalities of heart, brain, lung, liver and kidney function; 8. No serious mental illness; 9. Ability to comply with the plan; 10. the toxic and side effects of any previous chemotherapy have recovered to ≤CTCAE 1 grade or baseline level, except for sensory neuropathy or alopecia with stable symptoms ≤CTCAE 2 grade.

Exclusion Criteria:

1. People who are allergic to the ingredients in Yangzhengxiaoji Capsule
2. Have undergone major surgery within 3 weeks before the start of the study, or have not recovered any surgical effects after surgery, or have received chemotherapy.
3. patients who are combined with other cancers;
4. Patients with severe heart, liver, kidney and hematopoietic diseases; 5 Patients with poor compliance cannot take drugs according to regulations.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of nausea | 3 cycles (each cycle is 28 days)
  all grade of nausea base on CTCAE V5.0

SECONDARY OUTCOMES:
Quality of life changes | 3 cycles (each cycle is 28 days)
  base on Functional Assessment of Cancer Therapy-Ovarian Symptom Index (FOSI) score
PFS rate, PFS, OS and overall response rate (ORR, Overall response rate) at 12, 18 and 24 months | up to 24 months
  PFS rate, PFS, OS and overall response rate (ORR, Overall response rate) at 12, 18 and 24 months in patients with advanced ovarian cancer maintained on chemotherapy combined with bevacizumab switched nilaparib

OTHER OUTCOMES:
Incidence of anemia, thrombocytopenia, and neutropenia | 3 cycles (each cycle is 28 days)
  Incidence of All Grade Anemia, Thrombocytopenia, Neutropenia within 3 Cycles (CTCAE V5.0)
Incidence of fatigue | 3 cycles (each cycle is 28 days)
  Incidence of All Grade Fatigue Over 3 Cycles (CTCAE V5.0)

CONTACTS AND LOCATIONS:
Overall Officials: Guonan Zhang, Principal Investigator — Sichuan Cancer Hospital and Research Institute
Locations (1):
- Sicchuan cancer hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Torre LA, Trabert B, DeSantis CE, Miller KD, Samimi G, Runowicz CD, Gaudet MM, Jemal A, Siegel RL. Ovarian cancer statistics, 2018. CA Cancer J Clin. 2018 Jul;68(4):284-296. doi: 10.3322/caac.21456. Epub 2018 May 29. PMID 29809280
- [Background] Lord CJ, Ashworth A. PARP inhibitors: Synthetic lethality in the clinic. Science. 2017 Mar 17;355(6330):1152-1158. doi: 10.1126/science.aam7344. Epub 2017 Mar 16. PMID 28302823
- [Background] Pujade-Lauraine E, Ledermann JA, Selle F, Gebski V, Penson RT, Oza AM, Korach J, Huzarski T, Poveda A, Pignata S, Friedlander M, Colombo N, Harter P, Fujiwara K, Ray-Coquard I, Banerjee S, Liu J, Lowe ES, Bloomfield R, Pautier P; SOLO2/ENGOT-Ov21 investigators. Olaparib tablets as maintenance therapy in patients with platinum-sensitive, relapsed ovarian cancer and a BRCA1/2 mutation (SOLO2/ENGOT-Ov21): a double-blind, randomised, placebo-controlled, phase 3 trial. Lancet Oncol. 2017 Sep;18(9):1274-1284. doi: 10.1016/S1470-2045(17)30469-2. Epub 2017 Jul 25. PMID 28754483
- [Background] Mirza MR, Monk BJ, Herrstedt J, Oza AM, Mahner S, Redondo A, Fabbro M, Ledermann JA, Lorusso D, Vergote I, Ben-Baruch NE, Marth C, Madry R, Christensen RD, Berek JS, Dorum A, Tinker AV, du Bois A, Gonzalez-Martin A, Follana P, Benigno B, Rosenberg P, Gilbert L, Rimel BJ, Buscema J, Balser JP, Agarwal S, Matulonis UA; ENGOT-OV16/NOVA Investigators. Niraparib Maintenance Therapy in Platinum-Sensitive, Recurrent Ovarian Cancer. N Engl J Med. 2016 Dec 1;375(22):2154-2164. doi: 10.1056/NEJMoa1611310. Epub 2016 Oct 7. PMID 27717299
- [Background] Berek JS, Matulonis UA, Peen U, Ghatage P, Mahner S, Redondo A, Lesoin A, Colombo N, Vergote I, Rosengarten O, Ledermann J, Pineda M, Ellard S, Sehouli J, Gonzalez-Martin A, Berton-Rigaud D, Madry R, Reinthaller A, Hazard S, Guo W, Mirza MR. Safety and dose modification for patients receiving niraparib. Ann Oncol. 2018 Aug 1;29(8):1784-1792. doi: 10.1093/annonc/mdy181. PMID 29767688
- [Background] Ramos-Esquivel A, Viquez-Jaikel A, Fernandez C. Potential Drug-Drug and Herb-Drug Interactions in Patients With Cancer: A Prospective Study of Medication Surveillance. J Oncol Pract. 2017 Jul;13(7):e613-e622. doi: 10.1200/JOP.2017.020859. Epub 2017 Jun 19. PMID 28628392
- [Background] Ye L, Jia Y, Ji KE, Sanders AJ, Xue K, Ji J, Mason MD, Jiang WG. Traditional Chinese medicine in the prevention and treatment of cancer and cancer metastasis. Oncol Lett. 2015 Sep;10(3):1240-1250. doi: 10.3892/ol.2015.3459. Epub 2015 Jul 6. PMID 26622657
- [Background] 薛侃,等.养正消积胶囊应用于恶性肿瘤及癌前病变治疗中安全性的Meta分析[J].中国肿瘤临床.2013,40(21):1318-1323.
- [Background] 曲金荣.养正消积胶囊对晚期肺鳞癌患者GP方案化疗后骨髓抑制的防治作用[J].临床合理用药.2019.12(5):62-64.
- [Background] 宋圆圆.养正消积胶囊对癌因性疲乏患者的影响[J].天津中医药大学学报.2016.35(4):238-241.